CLINICAL TRIAL: NCT01349413
Title: Role of Gastroesophageal Acid Reflux at Squamo-columnar Junction in Functional Dyspepsia
Brief Title: BRAVO Study for Functional Dyspepsia
Acronym: BD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Justin Che-Yuen Wu, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: BD
Record Dates: First submitted 2011-05-05; First posted 2011-05-06 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Dyspepsia; Gastroesophageal Reflux
Keywords: Functional dyspepsia; symptom response; postprandial fullness; gastroesophageal reflux disease; acid suppression
MeSH Terms: conditions — Dyspepsia; Gastroesophageal Reflux | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Placebo (Placebo Comparator): Identical looking placebo (once daily)
  Interventions: Other: Placebo
- Esomeprazole 20mg daily (Experimental): Esomeprazole 20mg daily Oral for 8 weeks
  Interventions: Drug: Esomeprazole 20mg

INTERVENTIONS:
Drug: Esomeprazole 20mg — Oral Esomeprazole 20mg daily for 8 weeks
  Other Names: Nexium
  Arms: Esomeprazole 20mg daily
Other: Placebo — Identical looking placebo
  Arms: Placebo

SUMMARY:
Background:

Functional dyspepsia is one of the commonest digestive disorders. The pathophysiology of functional dyspepsia is uncertain. Proton pump inhibitor (PPI) has been recommended as the first line treatment for functional dyspepsia. However, the results on effectiveness of PPI are conflicting and it has been suggested that PPI is only effective for acid-related symptoms.

The investigators plan to use a wireless pH monitoring system positioned at the junction of esophagus and stomach to evaluate the chronological relationship between acid exposure at this region and symptoms of dyspepsia as well as its impact on the efficacy of acid suppressive therapy in treatment of functional dyspepsia.

Indication:

Functional dyspepsia patients

Study center(s):

Prince of Wales Hospital, Hong Kong

Aims:

1. To evaluate the chronological relationship between acid exposure at squamo-columnar junction (SCJ) and dyspeptic symptom in different subtypes of functional dyspepsia
2. To evaluate the relationship between acid exposure at squamo-columnar junction and dyspeptic symptom response to PPI
3. To compare the efficacy of PPI and placebo in treating functional dyspepsia patients

Study medication:

Esomeprazole 20mg vs Placebo o.d.

Study design:

Double-blind randomized placebo-controlled trial

Number of subjects: 130

Patient population:

Functional dyspepsia patients without concomitant gastroesophageal reflux disease (GERD)

Duration of study:

1 June 2010 - 30 May 2012

Primary variable(s):

Proportion of patients who report positive response to adequate relief of dyspeptic symptoms at week 8

Secondary variable(s):

Dyspeptic symptom scores, symptom association probability of dyspeptic symptoms in relation to esophageal pH of less than 4 as measured at 1 cm above SCJ.

Number of visits: 2

Hypothesis:

Increased acid exposure at SCJ contributes to dyspeptic symptom and predicts treatment response to PPI in FD patients without concomitant GERD

DETAILED DESCRIPTION:
Baseline assessment:

All patients will be invited to complete self-administered questionnaires for demographics and baseline symptom assessment

* Demographics: age, gender
* Screening of functional gastrointestinal disorder based on the Rome III questionnaires
* Functional dyspepsia symptom questionnaire: an 8-item dyspeptic symptom score questionnaire using 4-point (0-3) Likert scale based on recall of the past 7 days for assessment of epigastric pain, epigastric burning, belching, bloating, postprandial fullness, early satiation, nausea and vomiting. Functional dyspepsia will be further classified into epigastric pain syndrome (EPS) and postprandial distress syndrome (PDS) according to the Rome III definitions.
* Global dyspeptic symptom assessment: a dichotomous patient-reported scale in which they are asked to give a response of either "Yes" or "No" to the inquiry "Do you have adequate relief of dyspeptic symptom over the last 7 days?"
* GERD symptom questionnaire: Patients will also be asked to report the frequency of heartburn or acid regurgitation over the last 3 months. Patients with frequency of reflux symptoms of more than twice per month are deemed to have concomitant GERD and they will be excluded from the study.
* Psychological disorder: Patient Health Questionnaire (PHQ) will be used for screening of concomitant psychological disorder such as depression and generalized anxiety disorder.

Upper endoscopy and BRAVO pH capsule insertion:

Upper endoscopy will be arranged within 2 weeks of baseline assessment in order to exclude organic pathology such as peptic ulcer, esophagitis and neoplasm. The position and morphology of gastroesophageal junction is assessed during withdrawal of endoscope after deflation of stomach at end-expiratory of the patient in left lateral body position. The morphology of gastroesophageal junction will be graded according to the "flap valve" concept. In order to avoid the confounding effect of gross anatomical disruption of gastroesophageal junction on acid exposure at SCJ, patients with grade IV disruption of gastroesophageal junction, which refers to patulous hiatus with axial displacement of SCJ, will be excluded.

After completion of endoscopy examination, the BRAVO delivery system will be passed orally into esophagus in the same body position. The endoscope is then reintroduced to facilitate positioning of the delivery system under direct visualization. The BRAVO pH capsule will be placed at 1 cm proximal to SCJ for monitoring of acid exposure at SCJ.

Recording of esophageal pH profile and symptoms:

The wireless esophageal pH monitoring will last for 48 hours. During the study period, the patients will be instructed to engage in their usual daily activities. The patients will be given a diary documenting meals, sleeping and dyspeptic symptoms. The patient has to return the Bravo data recorder after 48 hours.

Randomization of treatment:

After completion of BRAVO pH monitoring, patients will be randomly assigned to either esomeprazole 20mg daily or identical looking placebo for 8 weeks. The random allocation sequence will be obtained from a computer-generated list of random numbers in blocks of 10. Concealed allocation is achieved by an independent staff who assigns treatments according to consecutive numbers in sealed envelopes. Study medications are dispensed as sealed packages in consecutive numbers. Medication adherence is measured by pill counts during final visit (V2).

Follow-up assessment:

The patients will report their individual dyspeptic symptoms on weekly basis using a self administered symptom questionnaire. At week 4 and week 8, they will need to give an additional rating on their overall symptom response using global symptom assessment. The patients are required to give a dichotomous response of either "yes" or "no" to the question stating "Do you have adequate relief of symptoms over the past 7 days?"

ELIGIBILITY:
Inclusion Criteria:

* Patients with functional dyspepsia that fulfill Rome III criteria with inadequate relief of dyspeptic symptoms
* Age >18
* Provision of written consent

Exclusion Criteria:

* Presence of organic pathology identified by upper endoscopy or other investigations
* Presence of sliding hiatus hernia as defined by flap valve grade IV disruption of morphology at gastro-esophageal junction
* Concurrent medications that affect gastrointestinal motility
* Presence of acid reflux or heartburn symptoms of more than twice a month
* History of gastric surgery
* H. pylori infection
* Use of PPI or NSAID in the past 4 weeks
* Pregnancy
* Known hypersensitivity to PPI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2011-08-24 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2018-07-19 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is the proportion of patients who report positive response to adequate relief of dyspeptic symptoms at week 8. | Week 8
  The proportion of patients who report positive response

SECONDARY OUTCOMES:
The secondary outcome measures include dyspeptic symptom scores, symptom association probability of dyspeptic symptoms in relation to esophageal pH of less than 4 as measured at 1 cm above SCJ. | 1st visit and 8 weeks
  Dyspeptic symptom scores, symptom association probability of dyspeptic symptoms in relation to esophageal pH

CONTACTS AND LOCATIONS:
Overall Officials: Justin CY Wu, MBChB(CUHK), Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Chinese University of Hong Kong — http://www.cuhk.edu.hk